CLINICAL TRIAL: NCT02743663
Title: The Development of Novel Clinical Tests to Diagnose and Monitor Asthma in Preschool Children
Acronym: WheezyER
Status: Completed | Type: Observational
Sponsor: The Hospital for Sick Children (Other)
Collaborators: Dalhousie University (Other)
Responsible Party: Principal Investigator, Padmaja Subbarao, Staff Respirologist, The Hospital for Sick Children
Other Study IDs: 1000041089
Record Dates: First submitted 2016-01-13; First posted 2016-04-19 (Estimated); Last update posted 2021-02-08 (Actual); Status verified 2021-02

CONDITIONS: Asthma; Wheeze; Obstructive Sleep Apnea; Food Allergy; Virus
Keywords: pediatric; lung ventilation inhomogeneity; preschool; asthma; wheeze
MeSH Terms: conditions — Asthma; Respiratory Sounds; Sleep Apnea, Obstructive; Food Hypersensitivity; Virus Diseases | interventions — Skin Tests; Albuterol; Blood Specimen Collection; Basophil Degranulation Test

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Venous blood samples collected and divided into DNA pellet, plasma, serum, and whole blood. Small portion of sample sent for Total IgE and CBC. The eosinophil and IgE information will be used to assist with categorizing wheezy subjects into API categories. The DNA sample will be analyzed using genome-wide association studies (GWAS), and looking for single-nucleotide polymorphism (SNPs) that are known to be associated with asthma. The whole blood samples will be used for the basophil activation test; Urine samples; Nasal swab samples; Nasal brush samples;
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Wheezing subjects: Two study visits will be completed with wheezing subjects. The baseline visit will be completed within a 5 day window from the child's discharge from the emergency department. The follow-up visit will be completed 3 months after the baseline visit. At both visits, participants will provide a nasal swab and urine sample, complete three breathing tests: multiple-breath washout, forced oscillation technique, and Spirometry. In addition, at the follow-up visit, children will have an allergy skin test done, a nasal brush to collect epithelial cells and provide a blood sample. Whole blood will be used for basophil activation test (BAT). Children age 4+ will also complete post-bronchodilator testing using Salbutamol to capture information about bronchodilator response.
  Interventions: Procedure: Bronchodilator response; Procedure: Allergy Skin Test; Procedure: Multiple-Breath Washout; Procedure: Forced Oscillation Technique; Procedure: Spirometry; Drug: salbutamol; Procedure: Nasal Brush; Procedure: Blood sample; Procedure: Basophil activation test; Procedure: Nasal swab
- Healthy cohort: One study visit will be completed with healthy participants. At this visit, three breathing tests will be performed: multiple-breath washout, forced oscillation technique, and spirometry. As well, an allergy skin test will be performed at the visit.
  Interventions: Procedure: Allergy Skin Test; Procedure: Multiple-Breath Washout; Procedure: Forced Oscillation Technique; Procedure: Spirometry

INTERVENTIONS:
Procedure: Bronchodilator response — Bronchodilator (Salbutamol - dose dependent on participant prescription) to wheezing subjects. 15 minutes after bronchodilator, spirometry and FOT repeated.
  Groups: Wheezing subjects
Procedure: Allergy Skin Test — Child will be tested for allergies to 17 different allergens, and positive (histamine) and negative (glycerin) controls, for a total of 19 allergens.
Procedure: Multiple-Breath Washout — Facemask in children 3-5 yrs, Wash-in phase: medical air inhaled during tidal breathing until steady state. Bias flow switched to 100% oxygen. Wash-out phase: patient breathes in 100% oxygen until nitrogen levels reach ~2%. Each test in duplicate and average is calculated.
  Other Names: MBW
Procedure: Forced Oscillation Technique — Sterile mouthpiece attached to FOT device. Patient is tested seated with noseclips and mouthpiece. FOT device produces oscillations at different frequencies (from that flow into lungs. Device measures resistance and reactance in lungs.
  Other Names: FOT
Procedure: Spirometry — Forced exhale manoeuvre completed by participant into flow meter, measuring forced exhale volumes and speed.
Drug: salbutamol — Given during bronchodilator response.
  Other Names: ventolin
  Groups: Wheezing subjects
Procedure: Nasal Brush — Nasal brush of 1 inferior turbinate to collect epithelial cells. Collected on either nare, choice dependent on how clear the nare is (i.e. no mucous, no nasal mucosal edema, no major structural impediments).
  Groups: Wheezing subjects
Procedure: Blood sample — 8mLs of venous blood collected using a butterfly needle of appropriate gauge. Blood sample used to collect CBC values, total IgE, serum, DNA, plasma, and whole blood.
  Groups: Wheezing subjects
Procedure: Basophil activation test — Collect basophils from whole blood sample, and expose cells to food allergens in flow cytometry machine to measure allergic response, if any.
  Other Names: BAT
  Groups: Wheezing subjects
Procedure: Nasal swab — Gentle swabbing of both nasal openings to collect mucous sample for analysis of microbial contents (i.e. bacteria, virus, fungi).
  Groups: Wheezing subjects

SUMMARY:
The study will ascertain the ability of preschool lung function tests to distinguish healthy children from those with wheeze, and to differentiate phenotypes of wheezy children (high and low risk for asthma as defined by API) in order to predict response to therapy, and to explore the correlation between preschool lung function test results and symptoms, in order to develop objective methods for monitoring asthma.

DETAILED DESCRIPTION:
In Canada, the most common chronic disease of childhood is asthma. Childhood asthma places a significant burden on the health care system (refn). No objective preschool asthma diagnostic tools exist, and the current gold-standard, the Asthma Predictive Index, does not provide information about lung function and symptom management. In this study, it is hypothesized that the lung clearance index (LCI), a value derived from the multiple breath washout test, will be the most sensitive, responsive discriminative test for preschool asthma. If it proves useful in the monitoring and diagnosis of preschool asthma, LCI has the potential to improve the clinical management and thus potentially significantly reduce hospitalization rates for preschool children suffering with asthma. In this unique data set, the investigators will also compare the relative utility of the forced oscillation technique (FOT) and preschool spirometry with the LCI in order to detect abnormalities amongst those children at high risk for preschool asthma. In addition, the impact of sleep apnea as a risk factor for and modifier of asthma will be investigated in this study. Furthermore, changes to the composition of the nasal microbiome during and after a wheezing episodes and the role of viral infections in wheezing exacerbations will be explored. Finally, the utility of new methods of diagnosing food allergy, such as the basophil activation test, will be examined in this Canadian cohort.

ELIGIBILITY:
Inclusion Criteria (Wheezing Subjects):

* 3 to 5 years of age (36 to 71 months)
* Diagnosis of Asthma made by a physician in the emergency department
* History of at least two other wheezing episode within the previous 12 months
* Received salbutamol within 4hrs before emergency department visit, during current emergency department visit, or was prescribed salbutamol at discharge from emergency department.

Inclusion Criteria (Healthy Controls):

* 3 to 5 years of age (36 to 71 months)
* Free of a respiratory infection for a minimum of 4 weeks prior to the testing visit

Exclusion Criteria (both subjects and controls):

* History or coexistence of renal, chronic pulmonary, cardiac, neurological or systemic disease
* Born pre-term (< 35 weeks GA)
* Insufficient command of the English language

Ages: 3 Years to 5 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Wheezing preschool-aged subjects will be recruited within 5 days of their discharge from the Emergency Department at the Hospital for Sick Children.
  Healthy preschool-aged controls will be recruited from the community (concurrent observational studies being conducted by the PI at the Hospital for Sick Children, children of co-workers)
Sampling Method: Non-Probability Sample
Enrollment: 121 (Actual)
Dates: Start 2014-06; Primary Completion 2020-12 (Actual); Study Completion 2020-12 (Actual)

PRIMARY OUTCOMES:
Change in Lung Clearance Index (LCI) in wheezing subjects. | baseline and 3 months
  Determine whether a change in LCI value captured over a 3 month period distinguishes two groups of wheezing children (high vs. low risk for asthma) as determined by the asthma predictive index (API).

SECONDARY OUTCOMES:
Obstructive Sleep Apnea (OSA) | Day 1, and again 3 months later.
  Obstructive sleep apnea symptoms in wheezing preschool aged children, captured using the Pediatric Sleep Questionnaire.
Change in asthma symptoms | baseline and 3 months
  Changes in parental report of symptoms (using the TRACK questionnaire) and clinically assessed symptoms (PRAM scale, ISAAC modified questions) over 3 month time frame.
Change in Forced Oscillation Technique (FOT) values in wheezing subjects. | baseline and 3 months
  Determine whether a change in FOT values (lung impedence) over 3 month period distinguishes two groups of wheezing children (high vs. low risk for asthma) as determined by API.
Change in spirometry values in wheezing subjects. | baseline and 3 months
  Determine whether a change in spirometric indices (i.e. FEV1, FEV0.75, FVC, FEV1/FVC,PEF) over a 3 month period distinguishes two groups of wheezing children (high vs. low risk for asthma) as determined by API.
Comparison of LCI values between wheezy subjects and healthy controls. | Day 1 for wheezing subjects and healthy controls, and again 3 months later for wheezing subjects.
  Determine if LCI values in preschool children differ between children with no history of wheeze and those with recurrent wheeze.
Comparison of forced oscillation technique (FOT; lung impedence) values between wheezy subjects and healthy controls. | Day 1 for wheezing subjects and healthy controls, and again 3 months later for wheezing subjects.
  Determine if FOT values in preschool children differ between children with no history of wheeze and those with recurrent wheeze.
Comparison of spirometric values between wheezy subjects and healthy controls. | Day 1 for wheezing subjects and healthy controls, and again 3 months later for wheezing subjects.
  Determine if spirometric indices (i.e. FEV1, FEV0.75, FVC, FEV1/FVC,PEF) in preschool children differ between children with no history of wheeze and those with recurrent wheeze.
Change in nasal microbiome in wheezing subjects | Day 1 and 3 months
  A nasal swab collected at Day 1 and again 3 months later will allow us to categorize the change in bacterial and viral communities of the nasal microbiome in wheezing subjects during and post wheezing exacerbations.
Viral infections causing wheezing | Day 1
  A nasal swab collected at Day 1 will be used to determine which viruses are causing wheezing in wheezing subjects.
Basophil activation test (BAT) | Day 1 and 3 months
  Determine the ability of the BAT to confirm food allergies in a wheezing cohort.
Lung epithelial cell immune response in wheezing subjects. | Day 1 and 3 months
  Epithelial lung cells collected from the inferior turbinate in wheezing subjects will be stimulated with viruses to categorize and differentiate immune cell response in wheezing subjects.

CONTACTS AND LOCATIONS:
Overall Officials: Padmaja Subbarao, MD, Principal Investigator — The Hospital for Sick Children
Locations (1):
- The Hospital for Sick Children, Toronto, Ontario, Canada